CLINICAL TRIAL: NCT04755621
Title: The Effect Of Core Stability Training on Pain, Function and Quality of Life in Individuals With Temporomandibular Disorders
Brief Title: The Effect Of Core Stability Training In Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Emre Serdar Atalay, Assist. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46418926-050.01.04
Record Dates: First submitted 2021-01-28; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Temporomandibular Disorder
Keywords: core stability; pain; quality of life; function; temporomandibular disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability Group (Experimental)
  Interventions: Other: Core stability training
- Control Group (Active Comparator)
  Interventions: Other: Rocabado Exercises

INTERVENTIONS:
Other: Core stability training — Core stability exercises
  Arms: Core stability Group
Other: Rocabado Exercises — Exercises for Temporomandibular Disorders
  Arms: Control Group

SUMMARY:
This study is to investigate the effect of Core stability training on pain, function, quality of life, sleep quality, body posture, foot posture, oral habits and kinesiophobia in individuals with temporomandibular disorder.

Materials and Methods: The study included 40 people over the age of 18, who were diagnosed with temporomandibular disorder from the dentist.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-55, diagnosed with temporomandibular disease by a dentist

Exclusion Criteria:

* Having received another treatment for TMR other than the use of night plate in the last 6 months
* Having a disease that can cause facial pain such as sinusitis, migraine, tension headache, trigeminal neuralgia
* Skeletal system fractures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Posture | 6 weeks
  New York Posture Scale
Sleep Quality | 6 weeks
  Pittsburg Sleep Quality Index
Kinesiophobia | 6 weeks
  Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK-TMD)
Oral Habits | 6 weeks
  Oral Behavior Checklist
Jaw Function | 6 weeks
  Jaw Functional Limitation Scale-20

SECONDARY OUTCOMES:
Foot Posture | 6 weeks
  Foot Posture Index-6
Graded Pain | 6 weeks
  Graded Chronic Pain Scale

CONTACTS AND LOCATIONS:
Overall Officials: Emre Serdar Atalay, PhD, Study Director — University of Health Sciences, Physical Therapy and Rehabilitation
Locations (1):
- University and Health Sciences Physical Therapy and Rehabilitation, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seyhan M, Atalay ES. Is core stability training effective in temporomandibular disorder? A randomized controlled trial. Clin Oral Investig. 2023 Dec;27(12):7237-7246. doi: 10.1007/s00784-023-05274-x. Epub 2023 Nov 4. PMID 37924356